CLINICAL TRIAL: NCT02581397
Title: Randomized Clinical Trial Evaluating the Non-clinical Inferiority of Suppository Transpulmin and Suppository Guaiacol Compared to Transpulmin Syrup in Frames of Productive Cough of Infectious Origin in Pediatric Participants.
Brief Title: Transpulmin Suppository and Guaiacol Compared to Transpulmin Syrup in Pediatric Participants With Productive Cough
Acronym: Transpulmin
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study stopped because after monitoring visits and data analysis we noticed a high number of protocol deviation that made impossible the results analysis.
Sponsor: Ache Laboratorios Farmaceuticos S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACH-TRN-03(01/10)
Record Dates: First submitted 2015-01-15; First posted 2015-10-21 (Estimated); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Cough
Keywords: cough; expectorant; upper respiratory tract infections; respiratory tract infections; antitussive agents
MeSH Terms: conditions — Cough; Respiratory Tract Infections | interventions — Guaiacol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Transpulmin suppository (Experimental): It is a rectal suppository that is manufactured by Aché S.A. and which is composed of camphor, eucalyptol, guaiacol and menthol.
  The rectal suppositories will be dispensed to 90 participants of this group within a cartridge. Each cartridge contains one strip with five suppositories.
  The participant must manage 1 suppository in the morning and 1 at night via rectal suppository (12/12h).
  The duration of treatment may be up to 03 or 07 days, depending on the visit discharge.
  Interventions: Drug: Transpulmin suppository
- Guaiacol suppository (Experimental): It is a rectal suppository that is manufactured by Aché S.A. and consists of guaiacol.
  The rectal suppositories will be dispensed to 90 participants of this group within a cartridge. Each cartridge contains one strip with five suppositories.
  The participant must manage 1 suppository in the morning and 1 at night via rectal suppository (12/12h).
  The duration of treatment may be up to 03 or 07 days, depending on the visit discharge.
  Interventions: Drug: Guaiacol suppository
- Transpulmin syrup (Active Comparator): It is a syrup which is manufactured by Aché S.A. and which is composed of guaifenesin.
  Transpulmin syrup will be dispensed to 90 participants of this group in a bottle of 150ml plus a dosing cup.
  The participant shall administer 7,5ml orally every 4 hours, The duration of treatment may be up to 07 days.
  Interventions: Drug: Transpulmin syrup

INTERVENTIONS:
Drug: Transpulmin suppository — 01 suppository in the morning and 01 at night, via rectal, for 03 or 07 days
  Other Names: Transpulmin
  Arms: Transpulmin suppository
Drug: Guaiacol suppository — 01 suppository in the morning and 01 at night, via rectal, for 03 or 07 days
  Other Names: Guaiacol
  Arms: Guaiacol suppository
Drug: Transpulmin syrup — 7,5ml every 4 hours, orally, for 03 or 07 days
  Other Names: Transpulmin
  Arms: Transpulmin syrup

SUMMARY:
This study evaluates the non-inferiority of Suppository Transpulmin and Suppository Guaiacol compared to Transpulmin Syrup in the treatment of cough with secretion of infectious origin in children between two and six years old. One third of participants will receive Suppository Transpulmin, the other one third will receive Suppository Guaiacol and the last one third will receive Transpulmin Syrup.

DETAILED DESCRIPTION:
Suppository Transpulmin, Suppository Guaiacol and Transpulmin Syrup are administered in the treatment of cough with secretion of infectious origin.

Each Suppository Transpulmin contains eucalyptol, menthol, camphor and guaiacol. The main pharmacological activity of eucalyptol occurs in the respiratory tract, playing expectorant action, fluidity and antiseptic. There are indications that eucalyptol be a controller inflammatory mediators, intervening directly in the pathophysiology of airway inflammation. On the other hand, menthol has spasmolytic effect antiflatulent, antipruritic, analgesic and antiemetic the mucosae, which has been shown in various studies in vitro and in vivo. In addition, effective against many kinds of bacteria and fungi. Camphor, in turn, is used in respiratory dysfunction due to secretolytic and antispasmodic properties (bronchi). Finally, the guaiacol is classified as an expectorant because it believes that promote increased sputum volume and decrease its viscosity, resulting in effective coughing. However, despite its extensive use in recent decades, there are few randomized controlled trials demonstrating its efficacy and tolerability, especially in pediatric participants.

Each Suppository Guaiacol contains guaiacol, whose action was explained previously.

Finally, each Transpulmin Syrup contains guaifenesin, which chemically it is a glyceryl ether guaiacol. Thus, their structures are similar, and their pharmacological effects and mechanisms of action. The addition of the hydroxyl group increases the hydrophilicity, making the compound more soluble, thus being more suitable for pharmaceutical syrup form.

ELIGIBILITY:
Inclusion Criteria:

* Participants and their guardians to accept the inclusion of the research participant in the study and agree to the terms proposed in the Informed Consent Form / Informed Assent Form, by signing the Informed Consent Form and Informed Assent Form by guardians and signature of Informed Assent Form by the participant, if possible;
* Participants aged ≥ (greater than or equal) to 02 years and ≤ (less than or equal) to 06 years, 11 months and 29 days of any ethnicity, class or social group;
* Participants diagnosed with acute respiratory disease of upper respiratory viral etiology (UAI) defined by medical researcher / sub-investigator, starting less than or equal to 48 hours prior to inclusion in the study;
* Participants with productive cough, sputum and lung snoring, so that the participant can be rated with a score of at least sporadic / light in specific score in accordance with paragraph 7.2.1. (Table 06 of the Protocol).

Exclusion Criteria:

* Participants treated with antibiotics;
* Clinical presence of bacterial infection of the upper airways and / or pulmonary (bacterial sinusitis, pneumonia, etc.);
* Participants with unproductive cough (dry cough);
* Treatment with immunosuppressants;
* Participating in the research that has participated in clinical trial protocols in the last twelve (12) months (National Board of Health- Resolution 251 of 07 August 1997, Part III, sub-item J), unless the investigator considers that there may be a direct benefit to it;
* Participants requiring multidrug treatment;
* Presence of other concomitant lung diseases that interfere, in the investigator's opinion on the study results;
* History hypersensitivity to components of the study drugs (suppository Transpulmin, Suppository of Guaiacol, Transpulmin syrup and Paracetamol);
* Subjects with pathologies that interfere with pulmonary function, such as cerebral palsy or muscular atrophies;
* Any medical or further processing (example: physiotherapy) that can interfere with the study objectives and / or participant safety;
* Participants with severe hepatic renal function disorders;
* Participants with x-ray chest compatible with bacterial infection framework;
* Participants with hemogram suggestive of bacterial infection;
* Medical history and / or changes in laboratory tests, clinical, physical and / or radiological that, judged by investigators, could compromise the participant's health or the reliability of data;
* Participants with previous diagnosis of diabetes mellitus type 01 or type 02;
* Participants diagnosed with porphyria;
* Participants who are in prohibited medication as described in item 6.9.1. of the Protocol.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 270 (Estimated)
Dates: Start 2015-05-05 (Actual); Primary Completion 2016-12-06 (Actual); Study Completion 2016-12-06 (Actual)

PRIMARY OUTCOMES:
Change of sputum, lung snoring, cough frequency and severity of coughing after three days (03 days ±1) of treatment. | (03 days ±1)
  The improvement of clinical signs and symptoms were evaluated for each parameter by using a 4-point rating scale: 0=none, 1=mild, 2=moderate, and 3=severe, after three days (03 days ±1) of treatment compared to baseline.

SECONDARY OUTCOMES:
Change of breathing difficulty, sleep quality, nasal obstruction, feeding and treatment adherence after three days (03 days ±1) of treatment. | (03 days ±1)
  The improvement of clinical signs and symptoms were evaluated for each parameter by using a 4-point rating scale: 0=none, 1=mild, 2=moderate, and 3=severe, after three days (03 days ±1) of treatment compared to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- L.A.L. Clínica Centro de Pesquisa e Desenvolvimento Ltda., Valinhos, São Paulo, Brazil